CLINICAL TRIAL: NCT02460939
Title: The Study on the Pulmonary Vessel Disease and Its Its Changes in Metabolism of Small Molecules
Brief Title: The Study on the Pulmonary Vessel Disease and Its Changes in Metabolism of Small Molecules
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Yingmin Ma, Vice president of the Beijing chaoyang hospital, Beijing Chao Yang Hospital
Other Study IDs: 12704102
Record Dates: First submitted 2015-06-01; First posted 2015-06-03 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Pulmonary Vessel Disease
Keywords: Pulmonary Vessel Disease; metabolism of small molecules

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to investigate the changes of the pulmonary vessel disease and its metabolism of small molecules.

DETAILED DESCRIPTION:
The patient with acute respiratory distress syndrome and sepsis come to hospital ,the investigators will blood them to study the changes in metabolism of small molecules.

ELIGIBILITY:
Inclusion Criteria:the aged between 18 and 85;Patients with ARDS and sepsis;Patients with only sepsis;normal

-

Exclusion Criteria:Age <18 or >85, pregnancy, diabetes mellitus, cardiac pulmonary edema, can lead to other conditions of ARDS: severe trauma, a large number of blood transfusions, severe acute pancreatitis, etc., end-stage tumor.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with ARDS and sepsis or only sepsis aged between 45 and 85
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-01 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
The changes of patients'metabolism of small molecules | about 10 days

CONTACTS AND LOCATIONS:
Overall Officials: yingmin ma, Study Director — Vice President of the Beijing chaoyang hospital
Locations (1):
- Liu Sijie, Beijing, Beijing Municipality, China